CLINICAL TRIAL: NCT00419237
Title: A Study to Investigate the Pharmacokinetics of a Single Inhaled Dose (400mcg) of GW685698X and Its Effect on Serum Cortisol in Patients With Impaired Liver Function and Matched Control Subjects.
Brief Title: Investigating The Pharmacokinetics Of An Inhaled Dose Of A New Corticosteroid In Patients With Impaired Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FFA10013
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Asthma
Keywords: hepatic impairment pharmacokinetics
MeSH Terms: conditions — Asthma

ARMS (2):
- Healthy subjects (Active Comparator): Subjects with normal liver function test will be administered a single oral inhaled dose of 400 micrograms (mcg) GW685698X in the morning of the study day. Each healthy subject will be matched as closely as possible for age, gender, bodyweight and race to a subject with impaired liver function.
  Interventions: Drug: GW685698X
- Subjects with hepatic impairment (Experimental): Subjects with Child Pugh B hepatic dysfunction will be administered a single oral inhaled dose of 400 mcg GW685698X in the morning of the study day.
  Interventions: Drug: GW685698X

INTERVENTIONS:
Drug: GW685698X — GW685698X will be available as dry white powder to be inhaled via DISKUS containing cellobiose octaacetate (COA) blended with lactose.

SUMMARY:
The proposed study is designed to investigate the pharmacokinetics, pharmacodynamics (as measured by serum cortisol) and safety of GW685698X in subjects with moderate hepatic impairment and in healthy subjects following a single oral inhaled dose of GW685698X. From the study results it should be possible to assess if there is an altered Risk: Benefit in patients with moderate hepatic impairment

ELIGIBILITY:
Inclusion:

* Are aged between 18-70 years, inclusive.
* If Female, you must be incapable of becoming pregnant.
* Show FEV1 of more than 70% of the predicted normal at screening.
* Are able to correctly use a DISKUS at the screening visit.
* Have Body Mass Index within the range of 19-33 kg/m2 inclusive.
* Do not show a positive pre-study urine drug screen.
* Do not show a positive pre-study blood alcohol test.
* Demonstrate a clinically normal 12-lead ECG at screening.
* Do not show a positive blood test for HIV.

If you are a Healthy Volunteer you must also:

* Have no significant abnormality on clinical examination.
* Have Liver Function Tests within the reference range at screening.

If you are a Patient Volunteer you must:

* Have moderate hepatic impairment
* Have no significant abnormality on clinical examination apart from hepatic impairment.

Exclusion:

* Suffered an upper respiratory infection in the 4 weeks before the screening visit.
* Suffered a lower respiratory infection in the 6 weeks before the screening visit.
* Taken oral corticosteroids in the 8 weeks before the screening visit.
* Taken inhaled, intranasal or topical steroids in the 4 weeks before the screening visit.
* A prolonged heartbeat (QTc interval >470msec).
* High blood pressure (systolic >160mmHg or diastolic >90mmHg) or as defined by the Investigator.
* Known sensitivity to corticosteroids.
* A history of lactose intolerance.
* A history of severe milk protein allergy.
* Donated blood in the last 3 months, or more than 1500mL (1000mL if female) in the last 12 months (including the amount taken for this study).
* Participated in a clinical trial within the last 3 months where you are/were exposed to a drug or device.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01-13 (Actual); Primary Completion 2005-04-15 (Actual); Study Completion 2005-04-15 (Actual)

PRIMARY OUTCOMES:
To investigate how impaired liver function affects the movement of single dose inhaled drug GW685698X within the body. Blood exposure levels in patients and matched control patients compared by taking blood samples after dosing | Up to Day 13

SECONDARY OUTCOMES:
Effect of GW685698X on serum cortisol by calculating weighted mean in blood over 24 hrs. Safety and tolerability of GW685698X in patients with impaired liver function from blood samples during dosing (clearance/distribution) and monitoring vital signs | Up to Day 13

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study FFA10013 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/FFA10013?search=study&search_terms=10013#rs
- Available data/document: Annotated Case Report Form: FFA10013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFA10013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFA10013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFA10013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFA10013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFA10013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFA10013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register